CLINICAL TRIAL: NCT03998709
Title: Effect of Fasting Free Fatty Acids and Fasting Glucose on 1st and 2nd Phase Insulin Secretion
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: results from other study suggest no good reason to proceed
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Adrian Vella, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-003325; R01DK078646 (NIH)
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Healthy
MeSH Terms: interventions — Somatostatin; Glucose; Insulin; Glucose Clamp Technique; soybean oil, phospholipid emulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elevation of fasting FFA and Glucose (Other): People with normal fasting glucose and normal fasting FFA (normal fasting glucose / normal glucose tolerance - NFG / NGT) will be studied on 2 occasions. On one occasion they will receive saline overnight and on the other they will receive intralipid and dextrose to raise fasting glucose and fasting FFA. Subsequently (on either study day) they will undergo a hyperglycemic clamp for 2 hours. After this somatostatin will be infused acutely to inhibit endogenous insulin secretion and observe clearance of beta-cell polypeptides.
  Interventions: Drug: Somatostatin; Other: Dextrose; Other: Intralipid
- Lowering of fasting FFA and glucose (Other): People with elevated fasting glucose and elevated fasting FFA (Impaired fasting glucose / impaired glucose tolerance - IFG / IGT) will be studied on 2 occasions. On one occasion they will receive saline overnight and on the other they will receive insulin to lower fasting glucose and fasting FFA. Subsequently (on either study day) they will undergo a hyperglycemic clamp for 2 hours. After this somatostatin will be infused acutely to inhibit endogenous insulin secretion and observe clearance of beta-cell polypeptides.
  Interventions: Drug: Somatostatin; Drug: Insulin

INTERVENTIONS:
Drug: Somatostatin — Somatostatin will be used to inhibit endogenous insulin secretion on either study day in both arms of the study
  Other Names: pancreatic clamp
Other: Dextrose — intravenous glucose will be used to raise fasting glucose in people with NFG / NGT
  Other Names: Elevation of glucose
  Arms: Elevation of fasting FFA and Glucose
Drug: Insulin — insulin will be used to lower fasting FFA and glucose in people with IFG / IGT
  Other Names: glucose clamp
  Arms: Lowering of fasting FFA and glucose
Other: Intralipid — intravenous intralipid (Fat Emulsion) will be used to raise fasting FFA in people with NFG / NGT
  Other Names: Elevation of FFA
  Arms: Elevation of fasting FFA and Glucose

SUMMARY:
Researchers are trying to determine how changes in fasting glucose and free fatty acids (products released from fat) affect insulin secretion.

DETAILED DESCRIPTION:
Non-invasive measurement of β-cell health is a long-hoped for tool in diabetes research. The observation that Type 2 Diabetes Mellitus (T2DM), and acute insulin resistance increase proinsulin concentrations led to the suggestion that a proinsulin/insulin ratio is a marker of β-cell integrity. However, proinsulin has a longer half-life (20-30min) than insulin (5min) and, unlike insulin, is not extracted by the liver. This limitation can only be overcome by direct and simultaneous measurement of insulin and proinsulin secretion. This experiment will measure in vivo proinsulin clearance so that proinsulin secretion can be calculated in people with differing degrees of glucose tolerance. It is also notable that subgroups of prediabetes differ in their fasting glucose and free fatty acid (FFA) concentrations. Whether short-term alteration of fasting glucose and FFA can alter subsequent prandial glucose metabolism is unknown. The loss of 1st phase insulin secretion(thought to represent release of pre-formed insulin granules) in T2DM can be partly restored by improved glycemic control although 2nd phase insulin secretion (thought to represent de novo synthesis of insulin) is unchanged. This experiment we will ascertain if changes in fasting FFA and glucose alter 1st and 2nd phase insulin secretion in people without diabetes.

ELIGIBILITY:
Inclusion Criteria

* Weight-stable, non-diabetic subjects from Biobank participants at Mayo Clinic, Rochester

Exclusion Criteria

* Age < 25 or > 65 years (to avoid studying subjects who could have latent type 1 diabetes, or the effects of age extremes in subjects with normal or impaired fasting glucose).
* HbA1c ≥ 6.5%
* Use of glucose-lowering agents.
* For female subjects: positive pregnancy test at the time of enrollment or study
* History of prior upper abdominal surgery such as adjustable gastric banding, pyloroplasty and vagotomy.
* Active systemic illness or malignancy.
* Symptomatic macrovascular or microvascular disease.
* Hormone replacement therapy >0.625 mg premarin daily

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
First phase of Insulin secretion in response to manipulation of fasting FFA and glucose | First 120 minutes of study
  1st phase of insulin secretion (Phi 1) - physiologic parameter
Second phase of Insulin secretion in response to manipulation of fasting FFA and glucose | First 120 minutes of study
  2nd phase of insulin secretion (Phi 2) - physiologic parameter

SECONDARY OUTCOMES:
proinsulin secretion in response to manipulation of fasting FFA and glucose | 2nd 120 minutes of the study
  proinsulin secretion - physiologic parameter
proinsulin clearance in response to manipulation of fasting FFA and glucose | 2nd 120 minutes of the study
  proinsulin clearance - physiologic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials